CLINICAL TRIAL: NCT07370116
Title: Safety and Feasibility of Omitting Nasogastric Decompression in Minimally Invasive Pancreaticoduodenectomy: a Multicenter Randomized Controlled Trial
Brief Title: Omitting Nasogastric Tube Decompression in Minimally Invasive Pancreaticoduodenectomy
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Collaborators: Zhejiang Provincial People's Hospital (Other); Shanghai Cancer Centre (Other); The Second Hospital of Hebei Medical University (Other); People's Hospital of Chongqing (Other); Shanghai Zhongshan Hospital (Other); Guangdong Provincial Hospital of Traditional Chinese Medicine (Other); Shandong Provincial Hospital (Other Government); The Second Affiliated Hospital of the Army Medical University (Unknown); West China Hospital (Other); Shanxi Province Cancer Hospital (Other)
Responsible Party: Principal Investigator, Min Wang, Professor; Chief Physician, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCC2025C1365
Record Dates: First submitted 2026-01-02; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Pancreaticoduodenectomy; Nasogastric Tube Decompression; Minimally Invasive Surgical Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- routine nasogastric tube (Active Comparator): standard nasogastric tube placement with the tube retained postoperatively
  Interventions: Procedure: nasogastric tube decompression
- routine omission of the nasogastric tube (Experimental): avoidance of prophylactic nasogastric tube placement
  Interventions: Procedure: Omission of nasogastric tube decompression

INTERVENTIONS:
Procedure: nasogastric tube decompression — Nasogastric tube decompression means standard NGT placement with the tube retained postoperatively until the drainage volume is <500 ml/day on postoperative day 3. Nasogastric tube placement will adhere to the following requirements: pre-insertion nasal patency assessment excluding the side with septal deviation or polyps, catheter pre-measurement from the apex nasi to the ear lobe and xiphoid process, and lubrication with liquid paraffin. After advancement into the pharynx, conscious patients will undergo repeated swallowing to facilitate passage, whereas unconscious patients will require laryngeal elevation with neck flexion to prevent tracheal intubation.
  Arms: routine nasogastric tube
Procedure: Omission of nasogastric tube decompression — Omission of nasogastric tube decompression means avoidance of prophylactic NGT placement throughout the perioperative period. If intraoperative NGT insertion becomes necessary because of acute gastric dilatation, the tube should be removed before anesthesia emergence.
  Arms: routine omission of the nasogastric tube

SUMMARY:
This study will evaluate two perioperative nasogastric tube strategies in patients undergoing laparoscopic pancreatoduodenectomy. The goal is to determine whether routine omission of a nasogastric tube is not worse than routine nasogastric tube placement in terms of overall complications and postoperative recovery.

Participants will be randomly assigned to one of two groups. Each group will receive the assigned nasogastric tube strategy during and after surgery, and will be followed during the hospital stay and after discharge for up to postoperative 90 days. Information will be collected from routine clinical care, including discomfort score, symptoms, imaging or laboratory tests when clinically indicated, and postoperative outcomes.

The main outcome of this study is the overall burden of postoperative complications within 30 days after surgery, measured using the Comprehensive Complication Index, which summarizes all complications into a single score. Secondary outcomes include rates of pancreas surgery-specific complications (such as delayed gastric emptying, pancreatic fistula, bile leak, bleeding, and chyle leak), other abdominal and pulmonary complications, and organ dysfunction (including kidney injury, sepsis, and new cardiac dysfunction). The study will also evaluate patient discomfort related to the nasogastric tube (pain/discomfort scores), the need for nasogastric tube reinsertion, postoperative recovery milestones (ability to resume oral intake and length of hospital stay), healthcare costs, and all-cause mortality at 30 and 90 days after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 years and 75 years.
2. Indication for MIPD confirmed by MDT evaluation.
3. Ability to understand trial requirements and willingness to adhere to study protocols.
4. Written informed consent obtained before registration.
5. Curative-intent treatment consistent with international clinical guidelines.

Exclusion Criteria:

1. Requirement of partial or total pancreatectomy or other palliative procedures, or presence of distant metastases (peritoneal, hepatic, distant nodal, or other organ involvement); therefore, these patients are not candidates for MIPD.
2. American Society of Anaesthesiologists (ASA) Physical Status ≥ IV.
3. Pregnant or breastfeeding women.
4. Severe psychiatric disorders.
5. History of other malignancy.
6. Neoadjuvant chemoradiotherapy prior to surgery.
7. Body mass index >35 kg/m2.
8. History of nasopharyngeal, gastric or oesophageal surgery.
9. Preoperative gastrointestinal obstruction.
10. Contraindications to nasogastric intubation, including recent caustic ingestion, oesophageal stricture/diverticulum, or maxillofacial trauma.
11. Participation in any other clinical trials within 3 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Comprehensive Complication Index | 30 days postoperatively
  Comprehensive Complication Index calculates a weighted sum of complications graded by the Clavien-Dindo classification that occur within 30 days postoperatively to generate a continuous score from 0 (no complications) to 100 (death), quantifying the overall postoperative complication burden

SECONDARY OUTCOMES:
pancreaticoduodenectomy-specific complications | 30 days postoperatively
  incidence of pancreaticoduodenectomy-specific complications, defined and classified according to International Study Group of Pancreatic Surgery criteria: delayed gastric emptying, postoperative pancreatic fistula, postoperative bile leak, postpancreatectomy haemorrhage, chyle leak and major complications (Clavien-Dindo grade ≥ II)
abdominal complications | 30 days postoperatively
  incidence of abdominal complications: surgical-site infection, intra-abdominal abscess, paralytic ileus, gastric dilatation and gastroenteric anastomotic leak
pulmonary complications | 30 days postoperatively
  incidence of pulmonary complications, including pneumonia, pulmonary embolism, atelectasis and pleural effusion
comfort | 30 days postoperatively
  nasogastric-tube-related discomfort scores (10-cm visual analogue scale)
Time to tolerate oral intake (liquids/solids) | Up to 90 days postoperatively
  Time from the end of surgery to the first time the participant begins and tolerates liquid (and separately solid) oral intake
Hospitalization cost | 90 days postoperatively
  Total hospitalization costs
Mortality rate | 90 days posoperatively
  all-cause mortality rate at postoperative 90 days
Rescue nasogastric tube insertion | 90 days postoperatively
  Postoperative placement (or reinsertion) of a nasogastric tube due to persistent distension, nausea, or vomiting, or if imaging was suggestive of gastrointestinal obstruction.
Length of stay | Up to 90 days postoperatively
  Days from the date of surgery to the date of discharge

CONTACTS AND LOCATIONS:
Overall Officials: Min Wang, Principal Investigator — Department of Pancreatic and Gastric Surgery, National Cancer Centre/National Clinical Research Centre for Cancer/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, China
Locations (1):
- National Cancer Center/National Clinical Research Center for Cancer/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data (IPD) underlying the results reported in publications, along with the data dictionary, will be made available.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Beginning 6 months after publication of the primary results and ending 5 years thereafter.
Access Criteria: Researchers who provide a methodologically sound proposal may request access. Proposals will be reviewed by the study team. Access will be provided after execution of a data use agreement. Data will be accessed via a secure platform or institutional controlled-access repository.